CLINICAL TRIAL: NCT00969696
Title: Galantamine Effects on Cognitive Function in Marijuana Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 0905005104; P50DA009241 (NIH); MIREC (Registry Identifier: Veteran's Administration)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Memory
Keywords: ability to learn, working memory
MeSH Terms: interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galatamine (Active Comparator): Galantamine is used for the treatment of mild to moderate Alzheimer's disease and various other memory
  Interventions: Drug: Galantamine
- Sugar Pill (Placebo Comparator): Sugar Pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 8Mg a day of a sugar pill
  Arms: Sugar Pill
Drug: Galantamine — 8mg of Galantamine
  Arms: Galatamine

SUMMARY:
To evaluate galantamine's effects on cognitive performance in marijuana users. Galantamine, an acetylcholine esterase inhibitor, is approved for treatment of Alzheimer's disease. Current marijuana users show impaired cognitive functioning, which predicts poor treatment response to behavioral treatments in this population. Whether cognitive impairment in marijuana users will improve with medication treatment has not been evaluated. We hypothesize that galantamine, compared to placebo, will improve cognitive performance in marijuana users.Galantamine, compared to placebo, will improve working memory, verbal learning/memory and response inhibition functions in marijuana users.

DETAILED DESCRIPTION:
To summarize, marijuana users show impaired cognitive functioning, especially in working memory and verbal learning and memory functions. Impaired cognitive functioning predicts poor treatment response in marijuana users. Whether the cognitive impairments in marijuana users improve with cholinergic enhancers has not been evaluated. In this double-blind, parallel-group study, we are proposing to evaluate galantamine's effects on cognitive performance in marijuana users. Thirty subjects will first have an adaptation session to familiarize them with the study procedures including cognitive assessment. The adaptation session will be followed by a 10-day treatment period, in which subjects will be randomized to galantamine (8 mg/day) or placebo. On Day 4 or 5 and Day 9 or10 of each treatment phase subjects will have test sessions, where a battery of cognitive tests will be administered. The cognitive test that will be administered will include the Hopkins Verbal Learning Test (HVLT) modules from the Cambridge Neuropsychological Test Automated Battery (CANTAB): the Rapid Visual Information Processing (RVIP) and the Stop Signal Test (SST).

Currently this study is in data analysis with 30 completers. (April 2011)

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 55 who are dependent on or abuse marijuana, according to DSM-IV criteria;
* History of marijuana use on the average of at least twice a week over a one-month period;
* Current marijuana use, indicated by positive urine toxicology for marijuana;
* No current medical problems and normal ECG;
* For women, neither pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* Current major psychiatric illnesses including mood, psychotic, or anxiety disorders;
* Current dependence to other drugs of abuse or alcohol (except nicotine or marijuana dependence);
* History of major medical illnesses including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal impairment and cardiac rhythm disturbances or other medical conditions that the study physician deems contraindicated for the subject to be in the study;
* Use of other medications including a) drugs that slow heart rate (eg, beta-blockers),which may increase the risk of bradycardia and AV block and b) NSAIDs; increased potential for developing ulcers/active or occult gastrointestinal bleeding;
* Known allergy to galantamine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
test whether galantamine in comparison to placebo, will improve cognitive functioning and the effects of galantamine on mood. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States